CLINICAL TRIAL: NCT00104338
Title: A Phase 2, Proof of Concept, Randomized, Open-label, Two-arm, Parallel Group, Multi-center Study to Assess the Efficacy and Safety of FK778 Compared With Standard Care in Renal Transplant Recipients With Untreated BK Nephropathy
Brief Title: Study of FK778 in Renal Transplant Recipients With Untreated BK Nephropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-0-196
Record Dates: First submitted 2005-02-24; First posted 2005-02-25 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: BK Polyomavirus; Kidney Diseases
Keywords: Investigational Therapies; Treatment Effectiveness; Treatment Efficacy; Immunosuppressant; BK Nephropathy; Polyomavirus, BK; Human Polyomavirus BK; Polyomavirus hominis 1
MeSH Terms: conditions — Kidney Diseases | interventions — 2-cyano-3-hydroxy-N-(4-(trifluoromethyl)phenyl)-2-hepten-6-ynamide

INTERVENTIONS:
Drug: FK778

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of a new oral immunosuppressant agent compared to standard care in renal transplant patients diagnosed with BK nephropathy.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of FK778 compared with standard care in renal transplant recipients with newly diagnosed and untreated BK nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipient with newly diagnosed BK nephropathy.

Exclusion Criteria:

* Previous treatment for BK nephropathy
* Organ transplant other than kidney
* Uncontrolled concomitant infection other than BK nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine BK viral load

SECONDARY OUTCOMES:
Change from baseline in plasma BK viral load
Change from baseline in renal function as measured by serum creatinine (SCr) and creatinine clearance (CrCl) at month 6 or at the end of therapy, whichever is earlier
Change from baseline in renal histology measured by Drachenberg criteria at month 6 or at the end of therapy, whichever is earlier

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Wichita, Kansas
  - Baltimore, Maryland
  - New Brunswick, New Jersey
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Harrisburg, Pennsylvania
  - Memphis, Tennessee
  - Salt Lake City, Utah
  - Fairfax, Virginia

REFERENCES:
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091